CLINICAL TRIAL: NCT06413836
Title: Effect of the Photodynamic Therapy Mediated by Methylene Blue in Surfactant Medium as an Adjuvant in the Treatment of Parts With Apical Periodontitis and the Presence of Fistula: A Randomized, Controlled Double-blind Clinical Trial
Brief Title: Evaluation of Photodynamic Therapy in Pieces With Presence of Fistula.
Acronym: aPDT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Renato Araujo Prates, Resercher, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCUUNINOVE
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Fistula
Keywords: Periodontitis; Fistula aPDT; Methylene Blue
MeSH Terms: conditions — Periodontitis; Fistula | interventions — Endodontics

STUDY DESIGN:
Intervention Model Description: Control Group (1): Mechanized endodontic treatment with CaOH (calcium hydroxide) medication between sessions. This medicine is the most commonly used in all conventional endodontic treatments.
  Study Group (2:) Mechanized endodontic treatment with CaOH (calcium hydroxide) medication following application of photodynamic therapy with methylene blue applied in surfactant medium.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will receive conventional endodontic treatment. The study group will receive antimicrobial photodynamic therapy with methylene blue application followed by active diode laser illumination. The control group will receive methylene blue solution and a simulation of laser application, which will be achieved by using an aluminum foil barrier placed at the tip of the equipment to block light in the control group. During this process, the participant will receive googles which aid eye protection and helps masking. The operator will wear protective glasses, which will aid in protection. Pre-irradiation and irradiation times will be the same at both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aPDT Therapy (Experimental): antimicrobial photodynamic therapy using methylene blue in surfactant solution
  Interventions: Device: aPDT; Procedure: Endodontic treatment
- conventional treatment (Sham Comparator): Endodontic treatment conventional treatment
  Interventions: Procedure: Endodontic treatment

INTERVENTIONS:
Device: aPDT — Mechanized endodontic treatment using an endodontic rotatory device (DENTSPLY) will be used to prepare the root canals. Following, it will be applied the methylene blue solution in surfactant medium and after 1 minute a diode laser equipment (DMC THERAPY/EC, Sao Carlos, Brazil) will be used to shine light at a wavelength of 660nm, 100 mW (miliWatts) and irradiation time of 3 min. CaOH (calcium hydroxide) paste will be applied at the root canals canals as a long-term dressing for endodontic treatment..
  Arms: aPDT Therapy
Procedure: Endodontic treatment — Mechanized endodontic treatment using an endodontic rotatory device (DENTSPLY) will be used to prepare the root canals. Following, it will be applied the methylene blue solution in surfactant medium and after 1 minute a diode laser equipment (DMC, THERAPY/EC, Sao Carlos, Brazil) will be used with an aluminium foil at the tip of the equipment to block light and use during 3 min as study group. CaOH (calcium hydroxide) will be applied at the root canals as a long-term dressing for endodontic treatment.

SUMMARY:
The goal of this clinical trial is to learn if adjuvant antimicrobial photodynamic therapy (aPDT) can help in the treatment in patients with pieces with apical periodontitis and the presence of fistula, in terms of reducing symptoms, resolution of fistula and the clinical signs of inflammation at the oral mucose, as well as, evaluation radiographic parameters.

Participants will undergo conventional endodontic treatment at Group I (n=15) and will undergo conventional endodontic treatment combined with antimicrobial photodynamic therapy at Group II(n=15).

DETAILED DESCRIPTION:
The calculation of the sample size was conducted with the statistical software G-Power 3.1 applying the chi-square homogeneity test. Identical sample sizes were considered for the aPDT group and the sham group. The percentage of type error was set at 5% and the statistical power at 80%, obtaining n = 30 considering 10% losses. The distribution of data within each group and the homogeneity of the variants will be verified for the choice of an analysis of variance or not. With this information the most proper statistical test will be conducted. The sample size calculation is based on the literature and a 5% significance level will be adopted

ELIGIBILITY:
Inclusion Criteria:

Patients must have a single-rooted tooth with apical periodontitis and the presence of fistula.

Patients must be over 18 years of age.

Exclusion Criteria:

Patients with comorbidities such as cancer, diabetes, coagulation diseases, and anemia; Patients undergoing orthodontic treatment; Patients with periodontal pockets deeper than 4 mm; Patients taking antibiotics; Pregnant or lactating patients; Patients with parts that present the impossibility of performing absolute isolation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fistula presence | Day 15
  Clinical observation to check presence or absence of fistula

SECONDARY OUTCOMES:
Radiographic register | Day 0 and Day 30
  Radiolucent radiograph analysis defining improvement or absence of improvement of the bone lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Prates, Study Director — University of Nove de Julho
Locations (1):
- UCU, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No